CLINICAL TRIAL: NCT03230539
Title: A proof-of Concept, Randomized 3-month Study to Evaluate the Effects of Three Contraceptive Intrauterine Systems Delivering Copper and a Daily Dose of 5, 20 or 40 μg of Ulipristal Acetate (UPA) on Ovulation, Endometrial Changes and Bleeding Patterns in Normally Cycling Women
Brief Title: A proof-of Concept, Randomized 3-month Study to Evaluate the Effects of Three Contraceptive Intrauterine Systems Delivering Copper and a Daily Dose of 5, 20 or 40 μg of Ulipristal Acetate (UPA)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Population Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 719
Record Dates: First submitted 2017-07-13; First posted 2017-07-26 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Contraception

STUDY DESIGN:
Intervention Model Description: A proof-of concept, randomized 3-month study to evaluate the effects of three contraceptive intrauterine systems delivering Copper and a daily dose of 5, 20 or 40 μg of Ulipristal Acetate (UPA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- UPA IUS 20 μg (Experimental): This is a proof-of-concept study utilizing a randomized dose-finding, parallel design to assess the effects of an IUS delivering Cu and 5, 20, or 40 μg of UPA over 12 weeks.
  Interventions: Drug: Ulipristal Acetate IUS delivering Cu and 20μg
- UPA IUS 5 μg (Experimental): This is a proof-of-concept study utilizing a randomized dose-finding, parallel design to assess the effects of an IUS delivering Cu and 5, 20, or 40 μg of UPA over 12 weeks
  Interventions: Drug: Ulipristal Acetate IUS delivering Cu and 5μg
- UPA IUS 40 μg (Experimental): This is a proof-of-concept study utilizing a randomized dose-finding, parallel design to assess the effects of an IUS delivering Cu and 5, 20, or 40 μg of UPA over 12 weeks
  Interventions: Drug: Ulipristal Acetate IUS delivering Cu and 40μg

INTERVENTIONS:
Drug: Ulipristal Acetate IUS delivering Cu and 5μg — This is a proof-of-concept study utilizing a randomized dose-finding, parallel design to assess the effects of an IUS delivering Cu and 5, 20, or 40 μg of UPA over 12 weeks.
  Arms: UPA IUS 5 μg
Drug: Ulipristal Acetate IUS delivering Cu and 20μg — This is a proof-of-concept study utilizing a randomized dose-finding, parallel design to assess the effects of an IUS delivering Cu and 5, 20, or 40 μg of UPA over 12 weeks.
  Arms: UPA IUS 20 μg
Drug: Ulipristal Acetate IUS delivering Cu and 40μg — This is a proof-of-concept study utilizing a randomized dose-finding, parallel design to assess the effects of an IUS delivering Cu and 5, 20, or 40 μg of UPA over 12 weeks.
  Arms: UPA IUS 40 μg

SUMMARY:
The UPA doses to be tested in this new IUS, 5, 20 or 40 μg per day, are not expected to suppress ovulation, however they should prevent endometrial growth resulting in endometrial atrophy, minimal bleeding, or even amenorrhea. It is anticipated that with low UPA doses, women will continue to ovulate and secrete progesterone (P) during the secretory phase of the menstrual cycle. As a result, PRM associated endometrial changes (PAECs) that have been described in previous UPA studies when ovulation was suppressed and associated with amenorrhea should not occur and endometria should retain normalcy. These expectations are based on our findings from a previous study in which the UPA doses tested were insufficient to block ovulation and participants maintained P secretion with normal endometria (protocol 349). Further evidence regarding the benefit of using low doses of UPA in a copper IUS stems from a small rhesus macaque proof of principle study that included an UPA-IUS delivering 40 or 60 μg/d of UPA, and fixed doses of E2 and cyclic P delivered via implants over 3 cycles.24 Indices of endometrial proliferation were significantly reduced in 3 out of 5 animals in that study; the endometria were atrophied with some glandular cysts, and typical PAECs were limited. Glands were generally small and tubular, however, in some animals they were large and dilated; resembling cysts with minimal evidence of proliferative activity.24 No bleeding was observed in the treated monkeys during progesterone withdrawal over the 3 cycles.

DETAILED DESCRIPTION:
Intrauterine devices (IUD) such as the Copper IUD (Paragard) and the levonorgestrel (LNG) IUS (Mirena®) are considered highly safe and effective long acting reversible methods of contraception (LARC). Nevertheless discontinuations are high due to user complaints of heavy bleeding during the first few months after insertion of IUDs or irregular bleeding in the first year of use of an IUS. To prevent these bleeding problems and enhance the overall safety profile, a new IUS is being developed that will deliver copper to provide its well described contraceptive efficacy in combination with UPA, a progesterone receptor modulator (PRM) that may decrease the amount of bleeding associated with use of a Cu IUD.

Since results of human studies delivering antiovulatory doses of UPA orally or with vaginal rings have shown endometrial changes characterized as typical PAECs, the occurrence of these endometrial effects with lower doses of the PRM delivered in the endometrium via this investigational IUS requires evaluation with both histology assessments and measures of proliferation markers. We need to determine if small doses of UPA administered locally with a new Cu-IUS with UPA can result in reduced bleeding or amenorrhea, as observed in the monkey study, and whether or not endometrial modifications occur.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women of reproductive age (21-38 years)
* Not at risk for pregnancy based on subject has undergone sterilization or subject is monogamous and her male partner has undergone sterilization
* Have regular menstrual cycles of 21-35 days duration
* Have an intact uterus and both ovaries
* Will be able to comply with the protocol
* Capable of giving informed consent

Exclusion Criteria:

* Women participating in another clinical trial within 30 days of initiation of this clinical trial
* Women not living in the catchment area of the clinic
* Known hypersensitivity to progestins or antiprogestins
* Known hypersensitivity to copper
* Any known chronic disease including HIV/AIDS
* All contraindications to IUD use,
* Desire to get pregnant during the study Breastfeeding
* Undiagnosed vaginal discharge or vaginal lesions or abnormalities
* Women with a current abnormal Pap. In accordance with the Bethesda system of classification: smear suggestive of high-grade pre-cancerous lesion(s), including HGSIL, are excluded;
* Women with LGSIL or ASCUS/high-risk HPV positive may participate if further evaluated with colposcopy and biopsy and no evidence of a lesion with a severity > CIN I is present and/or endocervical curettage is negative.
* Women with a biopsy finding of CIN I should have follow up for this finding per standard of care; women are excluded it treatment is indicated.
* Known benign or malignant liver tumors; known active liver disease
* Cancer (past history of any carcinoma or sarcoma)
* Medically diagnosed severe depression currently or in the past
* Known or suspected alcoholism or drug abuse
* Abnormal, clinically significant, serum fasting clinical chemistry values
* Women with known abnormal thyroid status
* Women with known impaired hypothalamic-pituitary-adrenal reserve
* Average diastolic BP > 85 mm or systolic BP >135 mm Hg after 5-10 minutes rest
* Body mass index (BMI) > 30.0 (or ≤18) Kg/m2
* Women with uterine anomalies
* Use within the past 2 months of any implanted hormonal contraceptives including progestin-releasing intrauterine systems (IUS) or progestin-releasing subdermal implants. NOTE: Removal of implanted hormonal contraceptives must have been for personal reasons unrelated to the purpose of enrollment in this study.
* Current use of a non-hormone containing IUD. NOTE: Removal of an IUD must be for personal reasons unrelated to the purpose of enrollment in this study.
* Use of injectable contraceptives during the previous 3 months (e.g. Cyclofem) or 6 months (e.g. DMPA).
* Women who do not have at least two progesterone measurements ≥10nmol/L during the baseline cycle will be excluded from further participation in the study (See Section 13.4.1)
* Acute pelvic inflammatory disease or a history of pelvic inflammatory disease unless there has been a subsequent intrauterine pregnancy. Postpartum endometritis or infected abortion in the past 3 months.
* Genital bleeding of unknown etiology.
* Untreated acute cervicitis or vaginitis, including bacterial vaginosis or other lower genital tract infections until infection is controlled.
* Current behavior suggesting a high risk for pelvic inflammatory disease
* Mucopurulent cervicitis
* Wilson's disease
* Allergy to any component of the IUS

Ages: 21 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the ability of the three doses of UPA as delivered by IUS to suppress bleeding. | 12 weeks
  Bleeding data obtained from diaries and CRFs.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Merkatz, RN, Study Director — Population Council
Locations (1):
- Profamilia, Santo Domingo, Dominican Republic